CLINICAL TRIAL: NCT05301907
Title: Survey Among Healthcare Professionals and MS Patients/Caregivers in Selected European Countries to Evaluate the Knowledge Required for the Safe Use of Mayzent
Brief Title: Survey Among Healthcare Professionals and MS Patients to Assess Their Understanding of RMP Materials
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CBAF312A2006; EUPAS44782 (Other: EU PAS number)
Record Dates: First submitted 2022-03-21; First posted 2022-03-31 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; MS; NIS; survey
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Health Care Professionals (HCPs): HCPs who prescribe, monitor and oversee the management / or provide in person medical supervision of patients on Mayzent (siponimod).
- Patients/Caregivers: Patients/Caregivers of patients who are taking Mayzent (siponimod) to treat their MS and according to the prescription of their neurologists across EU countries and Canada that were included in the launch program

SUMMARY:
Survey to be completed independently by HCPs (neurologists treating patients with MS and MS specialist nurses) and patients/caregivers.

DETAILED DESCRIPTION:
The survey- based study was conducting amongst HCPs and patients/caregivers in selected European countries including Germany, Netherlands, Nordics (Denmark, Sweden), Spain and Croatia, plus Canada, to evaluate whether HCPs and patients/caregivers receive the educational materials and to capture their knowledge of specific Mayzent (siponimod) safety measures.

ELIGIBILITY:
Inclusion Criteria:

Physicians were considered eligible for the survey if they meet the following screening criteria:

* Care for relapsing MS (RMS) patients
* Personally prescribed disease modifying therapies to MS patients, and;
* Have prescribed Mayzent (siponimod) in at least 1 SPMS patient.

Nurses were considered eligible for the survey if they:

* Provide supportive care for RMS patients
* Have initiated and/or managed the use of Mayzent (siponimod) in at least 1 SPMS patient.

Patient inclusion criteria include:

- Had initiated onto Mayzent (siponimod) to treat their MS since reimbursement

Exclusion Criteria:

-

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HCPs who prescribe, monitor and oversee the management / or provide in person medical supervision of patients on Mayzent (siponimod). And Patients/Caregivers of patients who are taking Mayzent (siponimod) to treat their MS and according to the prescription of their neurologists in selected EU countries
Sampling Method: Non-Probability Sample
Enrollment: 335 (Actual)
Dates: Start 2021-12-02 (Actual); Primary Completion 2025-05-16 (Actual); Study Completion 2025-05-16 (Actual)

PRIMARY OUTCOMES:
Percentage of HCPs and patients/caregivers who report receive and reading of the educational materials. | Throughout study completion, an average of 3 years
  Percentage of HCPs and patients/caregivers who report receive and reading of the educational materials to be collected
Knowledge and understanding of the HCPs as per detailed in the educational information provided | Throughout study completion, an average of 3 years
  Knowledge and understanding of the HCPs as per detailed in the educational information provided relating to:
  * The appropriate initiation
  * Specific safety measures when treating patients with Mayzent (siponimod)
  * Steps when treating patients with sinus bradycardia, 1st/2nd degree AV block or history of myocardial infarction or health failure
  * Procedures for the management of infections, macular edema, skin malignancies and pregnancy considerations.
  * Steps in ophthalmology checklist, managing infection risk, pregnancy, liver function and skin examinations
  Knowledge and understanding was measured according to the percentage of correct responses given across the sample, where 70% achieving the correct answer is deemed acceptable.
Knowledge and understanding of the patient/caregivers' as per detailed in the educational information provided | Throughout study completion, an average of 3 years
  Knowledge and understanding of the patient/caregivers' as per detailed in the educational information provided relating to:
  * Specific safety measures when being treated with Mayzent (siponimod)
  * Side effects and potential risks
  Knowledge and understanding was measured according to the percentage of correct responses given across the sample, where 70% achieving the correct answer is deemed acceptable.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Link to study results — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=18394